CLINICAL TRIAL: NCT01720238
Title: Clinical Effects and Cost-effectiveness Analysis of Early Anti-viral Therapy on HBV-related Compensated Liver Cirrhosis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Beijing Friendship Hospital (Other)
Collaborators: Peking University First Hospital (Other); Peking University People's Hospital (Other); Beijing YouAn Hospital (Other); Beijing Tiantan Hospital (Other); Beijing Ditan Hospital (Other); Peking Union Medical College Hospital (Other); Beijing 302 Hospital (Other)
Responsible Party: Principal Investigator, Jia Ji-Dong, Director of Liver Research Center, Beijing Friendship Hospital
Other Study IDs: D1211000039120003
Record Dates: First submitted 2012-10-31; First posted 2012-11-02 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2015-07

CONDITIONS: Liver Cirrhosis; Hepatitis B
Keywords: Compensated Liver Cirrhosis; Early Antiviral Therapy; Cost Effectiveness
MeSH Terms: conditions — Liver Cirrhosis; Hepatitis B | interventions — entecavir; Lamivudine; adefovir dipivoxil

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum,plasma and DNA
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Group 1: Entecavir Therapy
  Interventions: Drug: Entecavir
- Group 2: Lamivudine plus Adefovir Dipivoxil Therapy
  Interventions: Drug: Lamivudine plus Adefovir Dipivoxil

INTERVENTIONS:
Drug: Entecavir — 0.5mg qd
  Other Names: Baraclude; other manufacturers
  Groups: Group 1
Drug: Lamivudine plus Adefovir Dipivoxil — Lamivudine:100mg qd Adefovir Dipivoxil:10mg qd
  Other Names: Heptodin; other manufactures
  Groups: Group 2

SUMMARY:
Though newly reported HBV infection and HBsAg prevalence in China have greatly decreased, patients who had been chronically infected with HBV, especially those with liver cirrhosis cause great burden on public health care. In view of economic development level, drug availability and lack of independent health economics evidence, the investigators are still unable to give specific guidelines for HBV related compensated liver cirrhosis in China. Therefore, the investigators aim to investigate clinical effects and cost-effectiveness of two early anti-viral therapy strategies on HBV related compensated liver cirrhosis through this prospective, open-label, multicenter and nonrandomized study.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent
* aged 18-70 years
* clinical diagnosis of compensated liver cirrhosis

  1. liver biopsy showing cirrhosis
  2. endoscopy: esophageal varices , exclusion of noncirrhotic portal hypertension
  3. if no biopsy or endoscopy ，should meet two of the four:

     * Imaging(US, CT or MRI, et al) showing Surface nodularity： Echogenecity （spleen pachydiameter > 4.0cm or> 5 costal region）

       * PLT < 100×10 < 9 >/L，no other interpretation

         * ALB < 35.0 g/L, or INR > 1.3, or CHE < 5.0KU/L

           * Liver stiffness measurement value > 12.4 kpa
* HBeAg(+)with HBVDNA > 10 < 3 > IU/mL or HBeAg(-) wtih HBVDNA > 102 IU/mL

Exclusion Criteria:

* patient with decompensated liver cirrhosis:presence of ascites, variceal hemorrhage,hepatic encephalopathy
* allergic to any ingredients of the drugs
* patient complicated with alcoholic liver disease, autoimmune liver disease, heretic liver disease, drug induced liver disease,nonalcoholic liver disease or other chronic liver disease.
* AFP > 100ng/ml or Cr > 1.5×ULN
* pregnant woman
* patient with severe disease or other organ failure
* patient with any tumors
* patient with sever mental disease.
* patients with any disease or condition which the investigator or treating physician feels would interfere with the trial or the safety of the subject

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: compensated HBV Related liver cirrhosis
Sampling Method: Non-Probability Sample
Enrollment: 621 (Actual)
Dates: Start 2012-03; Primary Completion 2015-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Decompensation rate of liver cirrhosis | 3 years
  presence of ascites, variceal hemorrhage, hepatic encephalopathy and HCC

SECONDARY OUTCOMES:
child-pugh score | 1,2 and 3 years
HBVDNA undetected | 1,2 and 3 years
liver elasticity | 1, 2, and 3 years
life quality score | 1, 2 and 3 years
cost-effectiveness | 1, 2 and 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Dong Ji Jia, Doctor, Principal Investigator — Beijing Friendship Hospital
Locations (8):
- China (8):
  - Beijing Friendship Hospital, Beijing, Beijing Municipality
  - Beijing 302 Hospital, Beijing, Beijing Municipality
  - Beijing Ditan Hospital, Beijing, Beijing Municipality
  - Beijing Tiantan Hospital, Beijing, Beijing Municipality
  - Beijing YouAn Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - PeKing University People's Hopital, Beijing, Beijing Municipality
  - The First Hospital of Peking University, Beijing, Beijing Municipality

REFERENCES:
- [Derived] Wu X, Zhou J, Sun Y, Ding H, Chen G, Xie W, Piao H, Xu X, Jiang W, Ma H, Ma A, Chen Y, Xu M, Cheng J, Xu Y, Meng T, Wang B, Chen S, Shi Y, Kong Y, Ou X, You H, Jia J. Prediction of liver-related events in patients with compensated HBV-induced cirrhosis receiving antiviral therapy. Hepatol Int. 2021 Feb;15(1):82-92. doi: 10.1007/s12072-020-10114-1. Epub 2021 Jan 18. PMID 33460002